CLINICAL TRIAL: NCT06491823
Title: Sensorimotor Basis of Speech Motor Learning and Retention
Brief Title: Speech Motor Learning and Retention (Aim 2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000037622_b; 1R01DC022097-01A1 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-07-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Speech
Keywords: Speech Motor Learning; Retention
MeSH Terms: conditions — Speech | interventions — Acclimatization

STUDY DESIGN:
Intervention Model Description: Healthy right-handed adults with normal hearing will be recruited in equal number from both sexes. All participants will be fluent English speakers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MEPs (M1) / altered auditory feedback / MEPs + retention tests at 24h (Experimental): Evoked potentials will be recorded from brain area M1 (motor cortex) in combination with a speech motor learning procedure known as adaptation to altered auditory feedback. Retention of learning will be tested 24h later along with additional evoked potential recordings.
  Interventions: Behavioral: Adaptation; Device: Motor evoked potentials
- AEPs (A1) / altered auditory feedback / AEPs + retention tests at 24h (Experimental): Evoked potentials will be recorded from brain area A1 (auditory cortex) in combination with a speech motor learning procedure known as adaptation to altered auditory feedback. Retention of learning will be tested 24h later along with additional evoked potential recordings.
  Interventions: Behavioral: Adaptation; Device: Auditory evoked potentials
- SEPs (S1) / altered auditory feedback / SEPs + retention tests at 24h (Experimental): Evoked potentials will be recorded from brain area S1 (somatosensory cortex) in combination with a speech motor learning procedure known as adaptation to altered auditory feedback. Retention of learning will be tested 24h later along with additional evoked potential recordings.
  Interventions: Behavioral: Adaptation; Device: Somatosensory evoked potentials
- MEPs (M1) / unaltered auditory feedback / MEPs + retention tests at 24h (Experimental): Evoked potentials will be recorded from brain area M1 (motor cortex) in combination with unaltered auditory feedback. Retention of learning will be tested 24h later along with additional evoked potential recordings.
  Interventions: Behavioral: Adaptation baseline; Device: Motor evoked potentials
- AEPs (A1) / unaltered auditory feedback / AEPs + retention tests at 24h (Experimental): Evoked potentials will be recorded from brain area A1 (auditory cortex) in combination with unaltered auditory feedback. Retention of learning will be tested 24h later along with additional evoked potential recordings.
  Interventions: Behavioral: Adaptation baseline; Device: Auditory evoked potentials
- SEPs (S1) / unaltered auditory feedback / SEPs + retention tests at 24h (Experimental): Evoked potentials will be recorded from brain area S1 (somatosensory cortex) in combination with unaltered auditory feedback. Retention of learning will be tested 24h later along with additional evoked potential recordings.
  Interventions: Behavioral: Adaptation baseline; Device: Somatosensory evoked potentials

INTERVENTIONS:
Behavioral: Adaptation — Auditory adaptation in speech
  Arms: AEPs (A1) / altered auditory feedback / AEPs + retention tests at 24h; MEPs (M1) / altered auditory feedback / MEPs + retention tests at 24h; SEPs (S1) / altered auditory feedback / SEPs + retention tests at 24h
Behavioral: Adaptation baseline — Auditory baseline in speech
  Arms: AEPs (A1) / unaltered auditory feedback / AEPs + retention tests at 24h; MEPs (M1) / unaltered auditory feedback / MEPs + retention tests at 24h; SEPs (S1) / unaltered auditory feedback / SEPs + retention tests at 24h
Device: Motor evoked potentials — motor evoked potentials will be obtained in each recording block
  Arms: MEPs (M1) / altered auditory feedback / MEPs + retention tests at 24h; MEPs (M1) / unaltered auditory feedback / MEPs + retention tests at 24h
Device: Auditory evoked potentials — auditory evoked potentials will be obtained in each recording block
  Arms: AEPs (A1) / altered auditory feedback / AEPs + retention tests at 24h; AEPs (A1) / unaltered auditory feedback / AEPs + retention tests at 24h
Device: Somatosensory evoked potentials — Somatosensry evoked potentials will be obtained in each recording block
  Arms: SEPs (S1) / altered auditory feedback / SEPs + retention tests at 24h; SEPs (S1) / unaltered auditory feedback / SEPs + retention tests at 24h

SUMMARY:
The overall goal of this research is to test a new model of speech motor learning, whose central hypothesis is that learning and retention are associated with plasticity not only in motor areas of the brain but in auditory and somatosensory regions as well. The strategy for the proposed research is to identify individual brain areas that contribute causally to retention by disrupting their activity with transcranial magnetic stimulation (TMS). Investigators will also use functional magnetic resonance imaging (fMRI) which will enable identification of circuit-level activity which predicts either learning or retention of new movements, and hence test the specific contributions of candidate sensory and motor zones. In other studies, investigators will record sensory and motor evoked potentials over the course of learning to determine the temporal order in which individual sensory and cortical motor regions contribute. The goal here is to identify brain areas in which learning-related plasticity occurs first and which among these areas predict subsequent learning.

DETAILED DESCRIPTION:
The focus of this registration is Aim 2. Specific Aim 2 assesses the temporal order in which plasticity occurs in cortical motor and sensory brain areas during speech motor learning. Plasticity is assessed using measures of cortical excitability. Specifically, auditory, somatosensory and motor evoked potentials are elicited using single pulse TMS (motor), pure tone bursts (auditory), and mentalis nerve stimulation (somatosensory). Tests of cortical excitability are interleaved with trials involving speech motor adaptation. Cortical excitability is also measured using these same measures 24 hours after learning to assess retention.

The Speech Motor Learning and Retention Master Protocol is NCT06467292.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speakers
* Right-handed
* Normal hearing
* No speech disorder or reading disability

Exclusion Criteria:

* Cardiac pacemaker
* Aneurysm clip
* Heart or Vascular clip
* Prosthetic valve
* Metal implants
* Metal in brain, skull, or spinal cord
* Implanted neurostimulator
* Medication infusion device
* Cochlear implant or tinnitus (ringing in ears)
* Personal and/or family history of epilepsy or other neurological disorders or history of head concussion
* Psychoactive medications
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Speech motor learning | Performance as measured at the end of learning (30 minute session)
  Audapter software will be used to alter the first and second formant frequencies of the spoken words and this is played back to subjects through headphones. Subjects will be tested both with unaltered feedback and with abruptly introduced frequency shifts.The change in the first (F1) and second format frequency (F2) values will be assessed using Praat.
Retention of learning | 24 hours after learning (re-test lasts 30 minutes)
  The retention of adaptation to altered auditory feedback (and relearning) will be quantified in terms of F1 and F2 frequency shifts (relative to pre-training baseline). Larger values indicate more complete relearning or retention.
Motor evoked potentials (MEPs) | Performance as measured at the end of learning (30 minute session)
  Motor evoked potentials (MEPs) using single-pulse TMS will be recorded using surface electromyography (EMG) to measure MEP peak-to-peak response
Somatosensory evoked potentials (SEPs) | Performance as measured at the end of learning (30 minute session)
  Electrical stimulation will be used to elicit somatosensory evoked potentials (SEPs). SEPs will be recorded using electroencephalogram (EEG) to measure the SEP response in the interval 20 to 25 ms following stimulation (N20-P25 response).
Auditory evoked potentials (AEPs) | Performance as measured at the end of learning (30 minute session)
  Acoustical stimulation will be used to elicit auditory evoked potentials (AEPs). AEPs will be recorded using electroencephalogram (EEG) to measure the AEP response in the interval between the first positive peak and first negative peak following stimulation (P1-N1 response).

CONTACTS AND LOCATIONS:
Overall Officials: David Ostry, Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No